CLINICAL TRIAL: NCT00405912
Title: St. John's Wort for Tobacco Cessation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Amit Sood, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06-002296
Record Dates: First submitted 2006-11-29; First posted 2006-11-30 (Estimated); Results first posted 2011-04-18 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Smoking; Nicotine Dependence
MeSH Terms: conditions — Smoking; Tobacco Use Disorder | interventions — Hypericum extract LI 160

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Placeo (Placebo Comparator): Placebo pill was identical in appearance to the active medication.
  Interventions: Drug: Placebo
- St. John's Wort-900 mg/day (Experimental): St. John's Wort - 300 mg tablets, 3 times a day.
  Interventions: Drug: St. John's Wort-900 mg/day
- St. John's Wort-1800 mg/day (Experimental): St. John's Wort - 600 mg 3 times per day
  Interventions: Drug: St. John's Wort-1800mg/day

INTERVENTIONS:
Drug: Placebo — Placebo (inactive drug) given 3 times per day
  Other Names: inactive drug
  Arms: Placeo
Drug: St. John's Wort-900 mg/day — St. John's Wort - 300 mg tables -3 times per day
  Other Names: St. John's Wort
  Arms: St. John's Wort-900 mg/day
Drug: St. John's Wort-1800mg/day — St. John's Wort - 600 mg tables - 3 times per day
  Other Names: SJW
  Arms: St. John's Wort-1800 mg/day

SUMMARY:
After a steady decline for the last 50 years, the prevalence of tobacco use in the United States has reached a plateau of approximately 23%. Currently available treatments among adults are expensive and not efficacious for all tobacco users. New pharmacologic agents need to be developed and tested to achieve the Healthy People 2010 goal of less than a 12% adult tobacco use prevalence.

Bupropion, an FDA approved agent for tobacco cessation, acts by inhibiting central synaptosomal reuptake of dopamine and norepinephrine. A widely used herbal antidepressant, St. John's Wort (SJW), shares a similar mechanism of action and is effective for treating mild to moderate depression. SJW is well tolerated, available over the counter, and is significantly less expensive than the established treatments for tobacco dependence.

To date, no prospective clinical trial evaluating the efficacy of SJW for the treatment of tobacco use has been published. We propose to evaluate the efficacy of SJW for increasing tobacco abstinence and decreasing nicotine withdrawal symptoms in a randomized, double-blind, placebo-controlled, three-arm, parallel group, dose-ranging clinical trial. Participants (N=120) will be randomly assigned to one of the three groups and will receive a twelve-week course of SJW 900 mg per day, 1800 mg per day, or a matching placebo.

This study is anticipated to provide the data needed to develop a larger randomized controlled clinical trial submitted through the R01 funding mechanism.

DETAILED DESCRIPTION:
Cigarette smoking is the single most important preventable cause of morbidity, mortality and excess health care costs in the United States. The prevalence of cigarette smoking among U.S. adults has declined from 42% in 1965 to 20.9% in 2004. However, the overall decline is not occurring at a rate that will meet national health objectives by 2010. Available pharmacotherapies for the treatment of tobacco dependence are not efficacious for all tobacco users and have an overall estimated efficacy of approximately 20% for long-term tobacco cessation. Thus, novel pharmacotherapies for tobacco cessation need to be explored.

Current smokers tend to be younger with less education and belong to a lower socioeconomic status. Tobacco cessation treatments are expensive and often not covered by Medicare, Medicaid, or third party-payers. Our goal is to evaluate novel, safe, acceptable, effective, and inexpensive therapies that will increase tobacco abstinence rates.

The United States Public Health Service (USPHS) guideline recommends nicotine replacement therapy and bupropion as first-line agents for the treatment of tobacco dependence. Bupropion acts by central dopamine and norepinephrine reuptake inhibition. St. John's Wort (SJW), a widely used herbal product to treat mild to moderate depression, shares a similar mechanism of action and is available as a tobacco cessation aid in a number of over-the-counter preparations. While currently approved pharmacotherapies for tobacco dependence cost between $120-$240 per month, SJW is relatively inexpensive ($15 per month) and is well-tolerated. At present, no randomized prospective study of St. John's Wort for tobacco cessation has been published.

We plan to test the efficacy of SJW for tobacco cessation in a randomized, double-blind, placebo-controlled, three-arm, parallel group, dose-ranging clinical trial. We will obtain preliminary data about the efficacy of two different oral doses of SJW for improving tobacco abstinence rates and decreasing symptoms of nicotine withdrawal. All subjects will receive a behavioral intervention during participation in the study. A total of 120 subjects will be recruited into the study and randomly allocated to one of the three groups (groups A, B, and C). Participants in group A will receive SJW 300-mg three times a day for twelve weeks while participants in group B will receive SJW 600-mg three times a day for twelve weeks. Participants in group C will receive a matching placebo for the same duration.

We will conduct this research through the Nicotine Research Program (NRP) at the Mayo Clinic in Rochester, Minnesota. We are uniquely situated for completing this research as more than 7,500 patients have been enrolled in over 75 clinical trials conducted through the NRP. We propose the following specific aims:

Primary Aims:

1. To obtain preliminary evidence of the effect of a 12-week course of SJW in two different oral doses of 300-mg three times a day or 600-mg three times a day compared to placebo on the 7-day point prevalence tobacco abstinence rates at end of treatment and six months in 120 smokers.

Hypothesis: Cigarette smokers who receive SJW in two different oral doses of 300-mg three times a day or 600-mg three times a day for 12 weeks will have higher 7-day point prevalence tobacco abstinence rates at end of treatment and six months compared to cigarette smokers receiving placebo.

Secondary Aim:

1. To obtain preliminary estimates of the effect of a 12-week course of SJW in two different oral doses of 300-mg three times a day or 600-mg three times a day compared to placebo on prolonged tobacco abstinence rates at six months.

Hypothesis: Cigarette smokers who receive SJW in two different oral doses of 300-mg three times a day or 600-mg three times a day for 12-weeks will have higher prolonged tobacco abstinence rates at six months compared to cigarette smokers receiving placebo.

This study is innovative in that we are testing a novel therapeutic agent for the treatment of tobacco use. At the completion of this study, we expect to have obtained preliminary evidence regarding the effect of two different doses of SJW on symptoms of nicotine withdrawal and tobacco abstinence. We will also collect information on adverse effects of SJW in tobacco users and obtain data to plan a larger Phase III clinical trial, if the results from this trial suggest a potential for efficacy.

ELIGIBILITY:
A total of 120 subjects will be recruited in the study. Subjects will be eligible to participate if they:

1. Are at least 18 years of age;
2. Smoked more than10 cigarettes/day for the past one year;
3. Willing to make a quit attempt;
4. Able to participate fully in all aspects of the study; and
5. Have been provided with, understand, and have signed the informed consent.

Individuals will be excluded from study participation if they:

1. Meet diagnostic criteria for current major depressive disorder or lifetime history of bipolar disorder or schizophrenia. Patients with mild or moderate depressive symptoms [Beck Depression Inventory, Second Edition ≤ 28], but who do not meet current diagnostic criteria for major depressive disorder, will be included;
2. Are currently (within past 30 days) using antipsychotics or antidepressants;
3. Are currently (in previous 30 days) using any treatments for tobacco dependence (i.e., behavioral therapy, nicotine replacement therapy, bupropion SR, clonidine, or nortriptyline);
4. Have used an investigational drug within the 30 days prior to enrolling in this study;
5. Have ever used an herbal product for tobacco cessation;
6. Have recent history (in the past 3 months) of alcohol abuse or dependence as assessed by the CAGE questionnaire and study investigators;
7. Have a recent history of drug abuse as assessed by the Drug Abuse Screening Test 20 (DAST-20) and physician interview;
8. Are pregnant, lactating, or of child bearing potential, likely to become pregnant during the medication phase and not willing to use a reliable form of contraception. Reliable forms of contraception include barrier (diaphragm or condom with spermicidal jelly), injections, intrauterine device [IUD], surgical sterilization and abstinence;
9. Have a history of any major cardiovascular events in the past 6 months including unstable angina, acute MI or coronary angioplasty;
10. Have clinically significant acute or chronic progressive or unstable neurologic, hepatic, renal, cardiovascular, respiratory or metabolic disease;
11. Are currently on medications interacting with St. John?s Wort including warfarin, antiretrovirals (particularly indinavir and nevirapine), cyclosporine and tacrolimus, digoxin, nifedipine and verapamil, theophylline, all serotonergic drugs (serotonin reuptake inhibitors, tricyclic antidepressants, tramadol, venlafaxine, tryptophan and buspirone), MAO inhibitors, oral contraceptives, anti-cancer agents including imatinib and irinotecan, migraine medications (sumatriptan and zolmitriptan), methadone, lithium, sibutramine, atorvastatin and simvastatin, midazolam, alprazolam, fexofenadine, omeprazole, and general anesthetics (fentanyl, propofol, and sevoflurane);
12. Have another household member or relative participating in the study;
13. Have a known allergy to St. John?s Wort;
14. Have a history of photosensitivity;
15. Are professional drivers or operators of heavy machinery; and
16. Are scheduled for a planned surgical procedure within five days of taking SJW.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2005-09; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Sood, M.D., MSc, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Sood A, Ebbert JO, Prasad K, Croghan IT, Bauer B, Schroeder DR. A randomized clinical trial of St. John's wort for smoking cessation. J Altern Complement Med. 2010 Jul;16(7):761-7. doi: 10.1089/acm.2009.0445. PMID 20590478
- [Derived] Hajizadeh A, Howes S, Theodoulou A, Klemperer E, Hartmann-Boyce J, Livingstone-Banks J, Lindson N. Antidepressants for smoking cessation. Cochrane Database Syst Rev. 2023 May 24;5(5):CD000031. doi: 10.1002/14651858.CD000031.pub6. PMID 37230961

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began on 06/01/2006 and completed on 11/08/2007. Interested subjects who passed a phone prescreen were seen at a medical clinic (Mayo Clinic in Rochester, MN and Franciscan Skemp Medical Center in Lacrosse, WI) for consenting and additional study procedures to determine eligibility.
Groups:
- Placebo: The placebo pill was identical in appearance to the active medication. Dosage consisted of 1 pill by mouth three times per day. The medication was stopped at the end of 12 weeks.
- St. John's Wort - 900 mg /Day: St. John's Wort at a dose of 300 mg by mouth three times per day. The medication was stopped at the end of 12 weeks.
- St. John's Wort - 1800 mg /Day: St. John's Wort was initiated at a dose of 300 mg by mouth three times a day. The dose was increased after the first week to the target doses of 600 mg three times a day. This dose was continued for the next 11 weeks. The medication was stopped at the end of 12 weeks.
Period: Overall Study
Arm/Group | Placebo | St. John's Wort - 900 mg /Day | St. John's Wort - 1800 mg /Day
Started | 39 | 40 | 39
Completed | 23 | 21 | 23
Not Completed | 16 | 19 | 16
Not completed — Withdrawal by Subject | 12 | 11 | 12
Not completed — Lost to Follow-up | 4 | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | St. John's Wort - 900 mg /Day | St. John's Wort - 1800 mg /Day | Total
Number analyzed (Participants) | 39 | 40 | 39 | 118
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 1 | 2
  Between 18 and 65 years | 38 | 38 | 38 | 114
  >=65 years | 1 | 1 | 0 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 39.4 (13.0) | 38.3 (11.9) | 35.0 (12.2) | 37.6 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 18 | 21 | 65
  Male | 13 | 22 | 18 | 53
cigarettes per day [Mean (Standard Deviation); unit: cigarettes per day] — Self Reported average number of cigarettes smoked per day in the preceding 6 months prior to study enrollment.
  cigarettes per day | 19.4 (7.3) | 19.1 (7.2) | 21.0 (5.2) | 19.8 (6.6)

OUTCOME MEASURES:

1. Secondary Outcome: Number of Subjects With Prolonged Abstinence From Tobacco
Description: tobacco abstience during the 12-week course of SJW in two different oral doses of 300-mg three times a day or 600-mg three times a day compared to placebo at six months.
Time Frame: 24 weeks after the start of medication
Measure: Number; unit: participants
Arm/Group | Placebo | St. John's Wort - 900 mg /Day | St. John's Wort - 1800 mg /Day
Number analyzed (Participants) | 39 | 40 | 39
participants | 0 | 1 | 2
Statistical Analysis 1: Comparison: Placebo vs St. John's Wort - 900 mg /Day; Data were compared between treatment groups using Fisher's exact test for binary outcomes; Test type: Superiority or Other; p = 0.51, Fisher Exact; 1-sided test
Statistical Analysis 2: Comparison: Placebo vs St. John's Wort - 1800 mg /Day; Data were compared between treatment groups using Fisher's exact test for binary outcomes; Test type: Superiority or Other; p = 0.25, Fisher Exact; 1-sided test

2. Primary Outcome: Biochemically Confirmed 7-day Point Prevalence Abstinence From Tobacco
Description: Point prevalence tobacco abstinence was adjudicated if the following conditions were met:(a) self-reported tobacco abstinence for the previous 7 days with a negative response to the question "Have you used any type of tobacco,even a puff, in the past 7 days?" and (b) Expired Carbon Monoxide equal or less then 8 parts per million.
Time Frame: 12 weeks following start of medication
Measure: Number; unit: participants
Arm/Group | Placebo | St. John's Wort - 900 mg /Day | St. John's Wort - 1800 mg /Day
Number analyzed (Participants) | 39 | 40 | 39
participants | 7 | 8 | 6
Statistical Analysis 1: Comparison: Placebo vs St. John's Wort - 900 mg /Day; Data were compared between treatment groups using Fisher's exact test for binary outcomes; Test type: Superiority or Other; p = 0.52, Fisher Exact; 1 sided test
Statistical Analysis 2: Comparison: Placebo vs St. John's Wort - 1800 mg /Day; Data were compared between treatment groups using Fisher's exact test for binary outcomes; Test type: Superiority or Other; p = 0.73, Fisher Exact; 1-sided test

ADVERSE EVENTS:
Arm/Group | Placebo | St. John's Wort - 900 mg /Day | St. John's Wort - 1800 mg /Day
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/40 | 0/39
Other Adverse Events (participants affected / at risk) | 6/39 | 9/40 | 5/39
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=39) | St. John's Wort - 900 mg /Day (N=40) | St. John's Wort - 1800 mg /Day (N=39)
abdominal bloating (Gastrointestinal disorders) | 0 | 0 | 1
anxiety (Psychiatric disorders) | 1 | 0 | 0
dizziness (General disorders) | 1 | 0 | 0
dry mouth (General disorders) | 0 | 0 | 1
erectile dysfunction (General disorders) | 0 | 0 | 1
fatigue (General disorders) | 1 | 1 | 1
headache (General disorders) | 1 | 0 | 1
increased anger (General disorders) | 0 | 1 | 0
increased sweating (General disorders) | 1 | 0 | 0
insomnia (General disorders) | 1 | 4 | 1
sleep disturbance (General disorders) | 0 | 2 | 0
sunburn (General disorders) | 0 | 1 | 0
trouble concentrating (General disorders) | 1 | 0 | 0
vivid dreams (General disorders) | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No